CLINICAL TRIAL: NCT01536535
Title: Multicenter Open-label Study Evaluating the Safety and Efficacy of Standardized Initial Therapy Using Either Mesalamine or Corticosteroids Then Mesalamine to Treat Children and Adolescents With Newly Diagnosed Ulcerative Colitis.
Brief Title: Predicting Response to Standardized Pediatric Colitis Therapy
Acronym: PROTECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U01DK095745-01 (NIH); 1U34DK090804 (NIH)
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; mesalamine; corticosteroids; PROTECT
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine; Adrenal Cortex Hormones; Prednisone; Colectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mild UC (Experimental): Mild = Initiated on mesalazine, or on oral CS with Pediatric Ulcerative Colitis Activity Index (PUCAI) < 45
  Patients can be treated with any of the therapies noted below:
  Mesalazine: doses is rounded to the nearest 500mg increment, maximum dose of 75 mg/kg/day Oral corticosteroids:1-1.5 mg/kg/day, rounded up to the nearest 5 mg value
  IV corticosteroids:
  Additional Therapies:
  Calcineurin inhibitor (cyclosporine, tacrolimus) or anti-Tumour Necrosis Factor alpha (TNFα) therapy: These therapies may also be instituted if in the judgment of the attending physician is needed.
  Immunomodulator or biologic therapy: thiopurine then dosing of azathioprine:2.5-3 mg/kg/day; 6-MP at 1-1.5 mg/kg/day Colectomy
  Interventions: Drug: Mesalazine; Drug: IV Corticosteroid; Drug: Oral Corticosteroids; Other: Additional Therapies; Procedure: Colectomy
- Moderate to Severe UC (Experimental): Moderate/Severe = Initiated on IV CS, or oral CS with PUCAI ≥45
  Patients can be treated with any of the therapies noted below:
  Mesalazine: doses is rounded to the nearest 500mg increment, maximum dose of 75 mg/kg/day Oral corticosteroids:1-1.5 mg/kg/day, rounded up to the nearest 5 mg value
  IV corticosteroids:
  Additional Therapies:
  Calcineurin inhibitor (cyclosporine, tacrolimus) or anti-TNFα therapy: These therapies may also be instituted if in the judgment of the attending physician is needed.
  Immunomodulator or biologic therapy: thiopurine then dosing of azathioprine:2.5-3 mg/kg/day; 6-Mercaptopurine (MP) at 1-1.5 mg/kg/day Colectomy
  Interventions: Drug: Mesalazine; Drug: IV Corticosteroid; Drug: Oral Corticosteroids; Other: Additional Therapies; Procedure: Colectomy

INTERVENTIONS:
Drug: Mesalazine — Mesalazine (Pentasa) comes in 500mg capsules, and doses will need to be rounded to the nearest 500mg increment, with a maximum dose of 76 mg/kg/day. The average dose for the pediatric population will be approximately 70 mg/kg/day. Patients will be allowed to escalate to the final dose over 4 days to minimize side-effects such as headache.
  Other Names: Pentasa
Drug: IV Corticosteroid — Treatment with IV Corticosteroid
  Other Names: Prednisone
Drug: Oral Corticosteroids — Treatment with oral corticosteroids
  Other Names: Prednisone
Other: Additional Therapies — Anti-TNFα, Calcineurin inhibitor, Immunomodulator
Procedure: Colectomy — Colectomy

SUMMARY:
This is a multi-center, open-label study to determine the safety and effectiveness (how well it works) of two standardized treatments called "mesalamine" (Pentasa®) and "prednisone" in children with newly diagnosed Ulcerative Colitis (UC). Standardized treatments are types of treatments agreed upon and used by many qualified doctors. The medications being used in this study are considered "standard of care". Currently the ways in which these medicines are used (doses, frequency of dosing) may vary from site to site. This study will determine response to a standardized way of giving these medicines.

This study will also identify biomarkers for ulcerative colitis. Biomarkers are things that doctors can find in blood, stool, or bowel tissue that indicate how much inflammation there is in the bowel, how the inflammation is produced, and whether the inflammation is responding to treatment. Collecting response and remission (free of symptoms) information on these standardized treatments and the "biomarkers" can possibly help doctors create a model, or plan to know which children with UC may respond quickly, or which children may develop complications.

DETAILED DESCRIPTION:
Ulcerative Colitis (UC) denotes a phenotype of chronic inflammatory bowel disease (IBD), where inflammation is localized to the colonic mucosa, and extends from the rectum proximally in varying extents. The disorder is thought to result from an inappropriate activation of the mucosal immune system by antigens derived from both the host epithelium and the enteric flora, in genetically susceptible individuals. UC is strikingly heterogeneous with respect to age of onset, anatomical extent and disease course, with some experiencing chronically active severe disease, while others have intermittent periods of clinical remission and disease exacerbation. Patients' therapeutic responses vary. The reasons underlying such variability are not well understood. Although it has been widely hypothesized that several genes may influence the development of UC, and modify its phenotypic expression and severity, to date there are few confirmed examples of such relationships.

It has been postulated that the 5-aminosalicylate drugs exert their anti-inflammatory effect locally at the intestinal mucosa. Mechanisms likely include inhibition of 5-lipoxygenase resulting in decreased production of leukotriene B4, scavenging of reactive oxygen metabolites, prevention of up-regulation of leukocyte adhesion molecules, and inhibition of Interleukin 1 (IL-1) synthesis. Though multiple studies have shown the efficacy of aminosalicylates in inducing and maintaining remission in adults with UC, there are few data in children.

Corticosteroids (CS) have been the mainstay of treatment of severe UC since efficacy was first demonstrated in the 1955 randomized controlled trial by Truelove and Witts. Recent practice guidelines developed in adults support their use because of rapid onset of action and significant efficacy though CS dependency is noted. Though no controlled data on their use have been reported in children they are frequently used in this population. A recent report from investigators leading the prospective Pediatric IBD Collaborative Research Group Registry described 97 subjects with a diagnosis of UC and a minimum of 1 year follow-up; 79% received CS. At diagnosis 81% of CS treated patients had moderate/severe disease, and 81% had pancolitis. Clinically inactive disease, determined by physician global assessment, was noted in 60% at 3 months following CS therapy, but by one year 45% were considered CS dependent despite the frequent use of immunomodulators (IM). Among those children with initially moderate to severe disease in clinical remission at 3 months, about two-thirds had stopped the CS by one year.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 4years and ≤17 years at initiation of therapy (achieved 4th birthday, not yet 18th)
* Weight ≥15 kg
* New diagnosis of ulcerative colitis established by standard clinical, endoscopic, and histologic features at the PROTECT study site
* Colitis extending beyond the rectosigmoid (Paris classification E2, E3, or E4)[144]. If a patient is seriously ill and the clinician does not advance the colonoscope beyond the sigmoid colon but the clinical condition of the patient highly suggests more extensive disease then that patient is eligible for study.
* Disease activity by PUCAI of ≥10 at diagnosis
* No therapy previously initiated to treat the newly diagnosed ulcerative colitis
* Stool culture negative for routine enteric pathogens (Salmonella, Shigella, Campylobacter, E. coli 0157:H7) and Clostridium difficile toxin. Recent successful treatment for Clostridium difficile does not exclude a patient if toxin now absent. However, the patient must be a minimum of 5 weeks from the time treatment was started at the time toxin is absent.
* Stool study negative for enteric parasites (ova and parasites)
* Parent/guardian consent and patient assent
* Ability to remain in follow-up for a minimum of one year from diagnosis
* Female patients of child bearing age must have a negative urine pregnancy test and practice acceptable contraception (e.g., abstinence, intramuscular or hormonal contraception, two barrier methods (e.g., condom, diaphragm, or spermicide), intrauterine device, verbal report of the partner with history of vasectomy, or be surgically sterile). All female patients of childbearing potential (post-menarche) will undergo urine pregnancy testing at screening and must not be lactating.

Exclusion Criteria:

* Clinical, endoscopic, radiologic, or histologic evidence suggesting Crohn's disease (CD) consistent with Paris and North American Society for Pediatric Gastroenterology, Hepatology and Nutrition (NASPGHAN) criteria [144, 145]
* A previous diagnosis of inflammatory bowel disease for which treatment was given
* Evidence of any active enteric infection at the time of study entry
* Use of any oral CS for non-gastrointestinal indication within the past 4 weeks (e.g., asthma). Use of inhaled CS does not exclude a patient.
* History of use of IM or anti-TNFα agent for other medical conditions (e.g., juvenile rheumatoid arthritis) within the past 6 months
* Use of Accutane within the past 4 weeks
* Use of any investigational drug within the past four weeks
* Use of any 5-aminosalicylate within the past 4 weeks
* Pregnancy
* Subjects with poorly controlled medical conditions (e.g. diabetes, congestive heart failure)
* Proctitis or proctosigmoiditis only (Paris classification E1) on colonoscopic evaluation
* Chronic renal disease (BUN and serum creatinine >1.5 times the upper normal limit)
* Hepatic disease (AST or Alkaline phosphatase (ALP) greater than 3 times the upper normal limit in the absence of concomitant liver disease associated with IBD following full evaluation)
* History of allergy or hypersensitivity to salicylates, aminosalicylates, or any component of the Pentasa capsule.
* History of coexisting chronic illness or evidence of significant organic or psychiatric disease on medical history or physical examination, which, in the Investigator's opinion, would prevent participation in the study
* History or presence of any condition causing malabsorption or an effect on gastrointestinal (GI) motility, or history of extensive small bowel resection (greater than half the length of the small intestine).
* The finding of Helicobacter pylori at the time of evaluation does not exclude the patient from the study. Whether to treat this patient for Helicobacter pylori and when will be left to the discretion of the site.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 431 (Actual)
Dates: Start 2012-07-10 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Hyams, MD, Principal Investigator — Connecticut Children's Medical Center; Lee Denson, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Sonia Davis, DrPH, Principal Investigator — Collaborative Studies Coordinating Center - UNC-CH
Locations (29):
- United States (26):
  - UCLA Medical Center, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Nemours Children's Clinic, Jacksonville, Florida
  - Emory Children's Center, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Children's Hospital, Indianapolis, Indiana
  - John Hopkins Children's Hospital, Baltimore, Maryland
  - Children's Hospital of Boston, Boston, Massachusetts
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Goryeb Children's Hospital / Atlantic Health, Morristown, New Jersey
  - Women and Children's Hospital of Buffalo, Buffalo, New York
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Mt Sinai Hospital, New York, New York
  - Morgan Stanley Children's Hospital, New York, New York
  - Golisano Children's Hospital SUNY Upstate Medical University, Syracuse, New York
  - University of North Carolina at Chapel HIll, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Hasbro Children's Hospital, Providence, Rhode Island
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas
  - Primary Children's Medical Center (University of Utah), Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared 6 months after the primary publication of the manuscript appears on line.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will be shared 6 months after the primary publication of the manuscript appears on line.
Access Criteria: NIH repository list serve to be determined

REFERENCES:
- [Result] Hyams JS, Davis S, Mack DR, Boyle B, Griffiths AM, LeLeiko NS, Sauer CG, Keljo DJ, Markowitz J, Baker SS, Rosh J, Baldassano RN, Patel A, Pfefferkorn M, Otley A, Heyman M, Noe J, Oliva-Hemker M, Rufo P, Strople J, Ziring D, Guthery SL, Sudel B, Benkov K, Wali P, Moulton D, Evans J, Kappelman MD, Marquis A, Sylvester FA, Collins MH, Venkateswaran S, Dubinsky M, Tangpricha V, Spada KL, Britt A, Saul B, Gotman N, Wang J, Serrano J, Kugathasan S, Walters T, Denson LA. Factors associated with early outcomes following standardised therapy in children with ulcerative colitis (PROTECT): a multicentre inception cohort study. Lancet Gastroenterol Hepatol. 2017 Dec;2(12):855-868. doi: 10.1016/S2468-1253(17)30252-2. Epub 2017 Sep 20. PMID 28939374
- [Derived] Carmody JK, Plevinsky J, Peugh JL, Denson LA, Hyams JS, Lobato D, LeLeiko NS, Hommel KA. Longitudinal non-adherence predicts treatment escalation in paediatric ulcerative colitis. Aliment Pharmacol Ther. 2019 Oct;50(8):911-918. doi: 10.1111/apt.15445. Epub 2019 Aug 2. PMID 31373712
- [Derived] Hyams JS, Davis Thomas S, Gotman N, Haberman Y, Karns R, Schirmer M, Mo A, Mack DR, Boyle B, Griffiths AM, LeLeiko NS, Sauer CG, Keljo DJ, Markowitz J, Baker SS, Rosh J, Baldassano RN, Patel A, Pfefferkorn M, Otley A, Heyman M, Noe J, Oliva-Hemker M, Rufo PA, Strople J, Ziring D, Guthery SL, Sudel B, Benkov K, Wali P, Moulton D, Evans J, Kappelman MD, Marquis MA, Sylvester FA, Collins MH, Venkateswaran S, Dubinsky M, Tangpricha V, Spada KL, Saul B, Wang J, Serrano J, Hommel K, Marigorta UM, Gibson G, Xavier RJ, Kugathasan S, Walters T, Denson LA. Clinical and biological predictors of response to standardised paediatric colitis therapy (PROTECT): a multicentre inception cohort study. Lancet. 2019 Apr 27;393(10182):1708-1720. doi: 10.1016/S0140-6736(18)32592-3. Epub 2019 Mar 29. PMID 30935734

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment and enrollment began in July 2012 and ended in April 2015. Final study visits were in April 2016 at which time all study patients had a minimum of one year follow up. Patients were recruited from 29 centers in the United States and Canada.
Pre-assignment Details: Participants were consented at diagnostic colonoscopy obtaining biological specimens (DNA, serum, rectal tissue, stool for microbiome). After diagnosis of Ulcerative Colitis, they began treatment dictated by initial disease severity and provider/patient choice. Three patients were untreated.
Groups:
- Mild UC Disease: Mild = Initiated on mesalazine, or on oral CS with Pediatric Ulcerative Colitis Activity Index (PUCAI) < 45
- Moderate to Severe UC: Moderate/Severe = Initiated on IV CS, or oral CS with PUCAI ≥45
Period: Overall Study
Arm/Group | Mild UC Disease | Moderate to Severe UC
Started | 178 | 250
Completed | 163 (Patients either completed week 52 visit or had early colectomy or had additional therapy.) | 237 (Patients either completed week 52 visit or had early colectomy or had additional therapy.)
Not Completed | 15 | 13
Not completed — Withdrawal by Subject | 10 | 5
Not completed — Lost to Follow-up | 4 | 6
Not completed — Physician Decision | 1 | 1
Not completed — Participant moved | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Mild UC: Mild = Initiated on mesalamine, or on oral CS with PUCAI < 45
- Total: Total of all reporting groups
Arm/Group | Mild UC | Moderate to Severe UC | Total
Number analyzed (Participants) | 178 | 250 | 428
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.6 (3.4) | 12.7 (3.2) | 12.7 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 124 | 212
  Male | 90 | 126 | 216
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Corticosteroid Free Remission (SFR)
Description: Week 52 CS-free remission: Number of participants with a PUCAI < 10 and no corticosteroids (CS) for 28 days without additional therapy or colectomy. Participants in both groups received corticosteroids, biologics, or colectomies, if symptomatic.
  The Pediatric Ulcerative Colitis Activity Index (PUCAI) is a non-invasive disease activity index. The index measures include abdominal pain, rectal bleeding, stool consistency, number of stools per 24 hours, nocturnal stools, and activity level. A total score less than 10 indicates remission, Mild disease activity is 10-30, Moderate 35-60, Severe disease activity 65-85.
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Mild UC: Mild = Initiated on mesalazine, or on oral CS with PUCAI < 45
Arm/Group | Mild UC | Moderate to Severe UC
Number analyzed (Participants) | 163 | 237
Participants | 80 | 70

2. Primary Outcome: Number of Participants Who Needed Additional Therapy or Colectomy
Description: Number of participants who needed additional therapy or colectomy. Additional therapy included Anti-Tumour Necrosis Factor alpha (TNFα), Calcineurin inhibitor, Immunomodulator
Time Frame: Within 52 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Mild UC Disease: Mild = Initiated on mesalazine, or on oral CS with PUCAI < 45
Arm/Group | Mild UC Disease | Moderate to Severe UC
Number analyzed (Participants) | 163 | 237
Participants | 46 | 151

3. Secondary Outcome: Number of Participants Receiving a Colectomy
Description: Number of participants who received a colectomy within 52 weeks
Time Frame: Within 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mild UC Disease | Moderate to Severe UC
Number analyzed (Participants) | 163 | 237
Participants | 2 | 23

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Baseline through to the 52 week visit.
Groups:
- Mild UC: Mild = Initiated on 5-Aminosalicylates (ASA) or on oral CS with PUCAI < 45
- Moderate to Severe UC: Moderate/Severe = Initiated on IV CS or oral CS with PUCAI ≥45
Arm/Group | Mild UC | Moderate to Severe UC
All-Cause Mortality (participants affected / at risk) | 0/178 | 0/250
Serious Adverse Events (participants affected / at risk) | 21/178 | 79/250
Other Adverse Events (participants affected / at risk) | 157/178 | 224/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mild UC (N=178) | Moderate to Severe UC (N=250)
Hospitalized for UC complications (Gastrointestinal disorders) | 17 | 69
Pancreatitus acute (Hepatobiliary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
Clostridium difficile colitis (Gastrointestinal disorders) | 1 | 0
Dehydration (General disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 0 | 1
Hypersensitivity to mesalamine severe headache and pleuritic chest pain (Immune system disorders) | 0 | 1
Intentional Overdose (Psychiatric disorders) | 0 | 1
Intestinal anastomosis (Gastrointestinal disorders) | 0 | 1
Syncope (General disorders) | 0 | 1
Vasculitic rash (Immune system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mild UC (N=178) | Moderate to Severe UC (N=250)
Abdominal Pain (Gastrointestinal disorders) | 56 | 71
Diarrhea (Gastrointestinal disorders) | 52 | 71
Headache (General disorders) | 21 | 23
Nausea (Gastrointestinal disorders) | 10 | 17
Vomiting (Gastrointestinal disorders) | 7 | 11
Dyspepsia (Gastrointestinal disorders) | 4 | 11
Rash (Skin and subcutaneous tissue disorders) | 3 | 4
Acne (Skin and subcutaneous tissue disorders) | 1 | 11
Clostridium difficile (Gastrointestinal disorders) | 2 | 3
Pancreatitis (Hepatobiliary disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-02): https://cdn.clinicaltrials.gov/large-docs/35/NCT01536535/Prot_SAP_000.pdf